CLINICAL TRIAL: NCT03380078
Title: Effectiveness of a Multi-Level Implementation Strategy for ASD Interventions
Brief Title: Translating Evidence-based Interventions for ASD: Multi-Level Implementation Strategy
Acronym: TEAMS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of California, San Diego (Other); University of California, Los Angeles (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 990914; R01MH1198101 (Other Grant/Funding Number: NIMH); RO1MH1195001 (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2017-11-27; First posted 2017-12-20 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Implementation Mechanism; Autism Spectrum Disorder; Children's Mental Health Services; School Services
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Intervention Model Description: We will use a randomized factorial dismantling design to examine the independent and combined effectiveness of the TEAMS modules. MH programs (AIM HI study) and School districts (CPRT study) from San Diego, Sacramento, and LA Counties will be randomized to one of four conditions (STANDARD EBI-specific training only (control condition); TIPS (Motivational Module); TLI (LOCI Implementation Leadership Module).
  The Extension Study will use a "scale-out" open pilot design to examine the impact of a team enhanced TLI on provider and child outcomes.
Who Masked: Outcomes Assessor
Masking Description: Coders assessing provider outcomes are masked from study condition and aims.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard (Active Comparator): Programs assigned to the Standard condition will receive standard EBI training only
  Interventions: Behavioral: Classroom Pivotal Response Teaching (CPRT); Behavioral: An Individualized Mental Health Intervention for ASD (AIM HI)
- TEAMS Leadership Institute (TLI) ONLY (Experimental): Programs assigned to the TLI ONLY condition will receive standard EBI training for providers and leaders will participate in TLI.
  Interventions: Behavioral: Teams Leadership Institute (TLI); Behavioral: Classroom Pivotal Response Teaching (CPRT); Behavioral: An Individualized Mental Health Intervention for ASD (AIM HI); Behavioral: Team-Enhanced Teams Leadership Institute (TLI)
- Motivational Enhancement (TIPS for Training) ONLY (Experimental): Programs assigned to the TIPS ONLY condition will receive enhanced TIPS EBI training for providers.
  Interventions: Behavioral: Motivational Enhancement (TIPS for Training); Behavioral: Classroom Pivotal Response Teaching (CPRT); Behavioral: An Individualized Mental Health Intervention for ASD (AIM HI)
- TIPS + TLI (Experimental): Programs assigned to the TIPS + TLI condition will receive TIPS EBI training for providers and leaders will participate in TLI
  Interventions: Behavioral: Teams Leadership Institute (TLI); Behavioral: Motivational Enhancement (TIPS for Training); Behavioral: Classroom Pivotal Response Teaching (CPRT); Behavioral: An Individualized Mental Health Intervention for ASD (AIM HI)

INTERVENTIONS:
Behavioral: Teams Leadership Institute (TLI) — TLI is training for leaders in how to improve implementation of evidence-based interventions in community settings. TLI includes 5 key components : 1. Assessment: The Implementation Leadership Scale (ILS) and Implementation Climate Scale (ICS) will be completed by first-level leaders participating in the intervention, his/her subordinates (i.e. providers) and executive leaders. 2. Initial Training: a 3-hour didactic and interactive session that includes training in implementation leadership Leaders will develop a plan for using specific implementation support strategies. 3. Coaching: Weekly, brief (15-30 min) coaching calls keep leaders on track with goals and plans. Coaching includes review of progress toward goals, updating plan based on emergent issues, and problem solving. 4. Follow up : At month 4, leaders attend a 2-hour booster session . 5. Graduation: TLI programs will have a group-based graduation for the leaders and provider trainees at EBI training completion.
  Arms: TEAMS Leadership Institute (TLI) ONLY; TIPS + TLI
Behavioral: Motivational Enhancement (TIPS for Training) — The TIPS module applies MI principles and strategies to address attitudinal barriers and improve engagement in training. I AIM HI and CPRT trainers (in the TIPS Conditions ) will incorporate MI during training and ongoing consultation/coaching with providers to increase provider engagement and problem solving throughout training: 1. Providers will receive a call designed to provide information about training and the intervention. 2. During the workshop, trainers will assess concerns about participating and will use reflective problem solving to address barriers . Trainers will work with the provider to develop a plan through the use of Planning Worksheets . 3. During each consultation , planning worksheets will be updated collaboratively with the provider. 4. Providers will receive a weekly motivational text to encourage on-going participation.
  Arms: Motivational Enhancement (TIPS for Training) ONLY; TIPS + TLI
Behavioral: Classroom Pivotal Response Teaching (CPRT) — CPRT is a naturalistic behavioral intervention adapted from pivotal response training (PRT) for use during classroom activities to target social, communication, behavior, and learning skills. CPRT is a manualized program with user-friendly materials for training, intervention planning and fidelity monitoring provided in printed and web-based formats. CPRT has an established training plan and the training curriculum that follows the manual. Training and coaching including standard EBI training is conducted by MA or postdoctoral level researchers with extensive training and experience with CPRT.
Behavioral: An Individualized Mental Health Intervention for ASD (AIM HI) — A package of well-established, evidence-based behavioral strategies designed to reduce challenging behaviors in children served in MH service settings. AIM HI is a manualized program with user-friendly materials for training, intervention planning and fidelity monitoring provided in printed and web-based formats. AIM HI is a package of evidence-based parent-mediated and child focused strategies, designed to reduce behavior problems in children with ASD ages 5 to 13 served in MH programs. AIM HI has an established training plan and the training curriculum follows the manual. Training and coaching is conducted by MA or postdoctoral level researchers with extensive training and experience with AIM HI.
Behavioral: Team-Enhanced Teams Leadership Institute (TLI) — TLI-2 enhances TLI training by (a) including additional team members important to EBI implementation (e.g., supervisors, support staff) and (b) including the team in the development of an implementation plan using a team charter process. TLI-2 includes 5 components : 1. Assessment: The Implementation Climate Scale (ICS) will be completed by team members, providers, and executive leaders. 2. Initial Training: a 3-hour didactic and interactive session that includes training for the implementation team in implementation climate and development of an implementation plan. 3. Coaching: Bi-monthly, brief (15-30 min) coaching calls keep the team on track with goals and plans. Coaching includes review of progress toward goals, updating plan based on emergent issues, and problem solving. 4. Follow up: At month 4, team members attend a 2-hour booster session . 5. Graduation: TLI-2 programs will have a group-based graduation for the leaders and provider trainees at EBI training completion.
  Arms: TEAMS Leadership Institute (TLI) ONLY

SUMMARY:
The purpose of this study is to test the effectiveness of the "Translating Evidence-based Interventions (EBI) for ASD: Multi-Level Implementation Strategy" (TEAMS) model on provider-level implementation outcomes when used to enhance provider training in two evidence-based interventions for children with autism spectrum disorder (ASD). The TEAMS- Leadership Institute (TLI) module includes training to program/school district leaders in implementation of EBI, and the TEAMS Individualized Provider Strategy for Training (TIPS) module applies Motivational Interviewing strategies to facilitate individual provider behavior change. TEAMS will be tested in combination with two clinical interventions in two community service setting contexts (1) AIM HI intervention in mental health programs and (2) CPRT intervention in schools. It is expected that the addition of TLI and / or TIPS will improve use of EBI by community providers.

DETAILED DESCRIPTION:
Overview of Collaborative R01. The investigators propose to conduct two, coordinated studies testing the impact of the "Translating Evidence-based Interventions for ASD: A Multi-Level Implementation Strategy" (TEAMS). TEAMS focuses on improving implementation leadership, organizational climate (Teams Leadership Institute; TLI), and provider attitudes and engagement (TEAMS Individualized Provider Strategy for Training; TIPS) in order to improve two key implementation outcomes - ASD evidence-based intervention (EBI) fidelity, and subsequent child outcomes. The TLI module applies the LOCI ("Leadership and Organizational Change for Implementation") strategies, and the TIPS module applies MI (Motivational Interviewing) strategies to facilitate individual leader and provider level behavior change. These studies will use a randomized Hybrid implementation/effectiveness, Type 3, trial. Study #1 (PI: L Brookman-Frazee/UCSD) will test the TEAMS model with An Individualized Mental Health Intervention for ASD (AIM HI) in publicly-funded mental health services. Study #2 (PI: A Stahmer/UC Davis) will test TEAMS with Classroom Pivotal Response Teaching (CPRT) in school settings.

The Collaborative R01 mechanism will advance implementation science by allowing the research team to: 1) obtain a sufficient sample size to isolate the impact of individual and combined modules targeting different change mechanisms (implementation leadership/climate, attitudes); examine change mechanisms as mediators of outcomes; and provider background and organizational structure as moderators of outcomes; 2) enhance generalizability by testing TEAMS in combination with two clinical EBI in two public service systems critical for children with ASD; and maximize the diversity of the target population. Each site has unique expertise in one of the two EBI to be tested. The PIs have a strong history of collaboration and a clear management plan.

The Centers for Disease Control (CDC) estimates that 1 in 68 children have ASD. Long term outcomes for this populations are poor and the annual cost in the US is estimated to be $268 billion. Research on the effectiveness of methods to scale up EBI in routine care is critical to meet this growing public health need. The efficacy of a growing number of ASD EBI has been established. Emerging data from AIM HI and CPRT studies support the overall effectiveness of ASD EBI for improving child outcomes only when providers complete training and deliver interventions with fidelity. Unfortunately, adoption and provider training outcomes, considered key implementation outcomes, are variable (e.g., up to 35% of providers in our studies either do not complete training or have poor fidelity). These findings are especially concerning given the link between fidelity and child outcomes and the rapid increase of large-scale usual care implementation of EBI with little attention to training completion or fidelity, even with well-established training and consultation methods. Therefore, testing methods of improving implementation outcomes is key to ensuring positive child-level outcomes when EBI are implemented in routine care.

AIM HI and CPRT data indicate that (1) implementation leadership/climate and (2) provider attitudes towards EBI are promising targets of implementation interventions. The roles of both factors have been indicated for broader patient populations and also in current AIM HI and CPRT projects. As such, the project will apply two, established interventions (LOCI, MI) in the TEAMS model to target these specific mechanisms of change. This study will test the impact of combining standard, EBI-specific training with the two TEAMS modules individually and together on multiple implementation outcomes. A dismantling design will be used to understand the effectiveness of TEAMS and the mechanisms of change across settings and participants. The specific aims and hypotheses are:

1. Test the effectiveness of the TEAMS modules individually and in combination on implementation outcomes when paired with two ASD EBI.

   a) Compared to standard ASD EBI training (control) and individual TEAMS modules (LEAD or PROV), the full TEAMS model will lead to more positive implementation outcomes for providers (training completion, fidelity), and children (improvements in targeted symptoms).
2. Test the impact of TEAMS modules on organization and provider level mechanisms of change.

   a) TEAMS-LEAD will increase use of implementation leadership strategies and TEAMS-PROV will lead to greater changes in provider attitudes and engagement in EBI training.
3. Identify moderators and mediators of implementation outcomes.

   1. Identify provider and organization characteristics that moderate implementation outcomes; and
   2. Identify provider and leader level mechanisms of change that mediate implementation outcomes.

Team Enhanced TLI Supplemental study Our supplemental study will examine whether a team-enhanced version of TLI results in better provider and child outcomes outcomes compared to TLI.

Impact: This implementation intervention has the potential to increase quality of care for ASD by improving effectiveness of EBI implementation. The process and modules will be generalizable to multiple service systems, providers, and interventions, providing broad impact in mental health, educational and community services.

ELIGIBILITY:
The combined multi-level sample for both studies will include 74 programs/districts, 148 agency/district leaders, 590 providers (average of 8 per program/district) and 590 parents (1 per provider). It is estimated that an additional 590 participants will complete the 360 Organizational Assessment. Providers are expected to be approximately 85% female and 35% Hispanic. Parent participants are expected to be approximately 80% female and 60% Hispanic.

Mental health programs will be those providing publicly funded psychotherapy services to children in San Diego, Sacramento and LA Counties for in person training and throughout California for distance training. Districts will be those providing public education services to elementary school children with ASD in San Diego, Sacramento and LA Counties for in person training and throughout California for distance training.

Inclusion Criteria for Leaders

(1) Identified as Program Managers at an enrolled site or identified as Program Specialist in an enrolled program/district

Inclusion Criteria for Providers

1. Employed at a participating program/district
2. Employed for at least the next 7 months
3. Has an eligible child on current caseload/classroom (see below)
4. Did not participate in the AIM HI or CPRT effectiveness studies

Inclusion Criteria for Parent Participants (enrolled in a dyad with participating provider)

1. Has a child age 3-13 years.
2. Has a child with a current ASD diagnosis on record or a primary educational classification of autism as indicated in school records

Inclusion Criteria for 360 degree Organizational Assessment

1. Identified as a leader or provider at enrolled site
2. Linked to a participant leader (either as a supervisor or direct report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1206 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Provider Training Completion / Certification | Certification will be determine at POST training (6 mos)
  Provider training/consultation completion will be measured through completion of requirements for certification, including attendance at workshops and training, completion of appropriate planning tools to program standards and meeting trainer rated fidelity of implementation standards.

SECONDARY OUTCOMES:
Child Improvements on The Eyberg Child Behavior Inventory (ECBI) | Child measures will be rated at PRE (intake) and POST intervention (6 mos)
  The ECBI is a 36 item paper-and-pencil rating scales completed by parents that assesses the severity of conduct problems in children as well as the extent to which parents find the behaviors troublesome. It assesses the frequency of disruptive behaviors occurring in the home setting. It provides an Intensity Raw Score and a Problem Raw Score. Internal consistency reliability (Cronbach's alpha): .95 for the Intensity scale and .93 for the Problem scale; (2) Test-retest reliability: .75 to .86 for the Intensity scale and .75 to .88 for the Problem scale; (3) Inter-rater reliability: .86 for the Intensity scale and .79 for the Problem scale.
Child Improvements on the PDD Behavior Inventory, Parent Extended Version (PDDBI-PX) | Child measures will be rated with the target child at PRE (intake) and POST intervention (6 mos)
  PDDBI-PX is a 188-item, paper-and-pencil rating scale completed by parents designed to assess symptoms of autism spectrum disorder and responsiveness to intervention in children. Subscales measure maladaptive (sensory/perceptual approach behaviors; fears; arousal problems; aggressiveness /behavior problems; social pragmatic problems) and adaptive behaviors (social approach; learning, memory and receptive language; phonological skills; pragmatic ability). Domain, composite, and total autism scores are provided. (1) Internal consistency reliability (Cronbach's alpha): ranged from .79 to .97 for all subscales; (2) Test-retest reliability: ranged from .38 to .91 over a 12-month interval; (3) Inter-rater reliability: Parent-Teacher ranged from .55-.67.

OTHER OUTCOMES:
Training/consultation attendance | Attendance will be tracked throughout intervention training and compiled at Post Intervention (6 months)
  Attendance will be tracked by trainers on a program developed form.
Evidence-Based Practice Attitude Scale (EBPAS-15) | Measures will be completed at PRE (intake) and POST intervention (6 mos)
  This measure includes the 15 items in the original Evidence-Based Practice Attitude Scale (EBPAS-15; Aarons, 2004; Aarons, Glisson, Hoagwood, et al., 2010). The EBPAS assesses provider attitudes toward adoption of EBP in public sector service settings and has been used in substance use disorder treatment, mental health, medical, and social service settings. The EBPAS consists of a higher-order factor/total scale (i.e., total scale score), representing respondents' global attitudes toward adoption of EBPs, and four lower-order factors/subscales. The EBPAS demonstrates good internal consistency reliability (α = .76) and concurrent and predictive validity. Supervisors and providers will complete this measure.
Implementation Leadership Scales | Measures will be completed at PRE (intake) and POST intervention (6 mos)
  The Implementation Leadership Scale (ILS; Aarons, Ehrhart, & Farahnak, 2014) includes four subscales that assess the degree to which a leader is knowledgeable, supportive, proactive, and perseverant in implementing EBP. The ILS demonstrates excellent internal consistency reliability (α = .98, 12 items) and convergent and discriminant validity. Providers will complete this measure about their supervisors and executives will complete the measure about the supervisors that they oversee. Each supervisor will also rate him/herself.
Implementation Climate Scales | Measures will be completed at PRE (intake) and POST intervention (6 mos)
  The Implementation Climate Scale (ICS) was originally developed as a part of an NIMH measure development grant (R21MH098124, PI: Ehrhart). This 18-item measure assesses the degree to which there is a strategic organizational climate supportive of evidence-based practice implementation. Implementation climate is defined as employees' shared perceptions of the policies, practices, procedures, and behaviors that are rewarded, supported, and expected in order to facilitate effective EBP implementation. The ICS demonstrates excellent internal consistency reliability (α = . 912, 18 items) and convergent and discriminant validity. Providers and supervisors will complete this measure.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California, Davis, Sacramento, California
  - University of California, San Diego, San Diego, California
  - University of California, Los Angeles, Westwood, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
1. Submit an NIMH Data Archive Data Submission Agreement and work with NDCT staff to develop a data submission schedule and outline data elements to be submitted. 2. Data collection will be carefully organized and documented following best practices for data file management to allow for data sharing. 3. Include appropriate language in subject consent documents to allow for the broad sharing of data through NDCT. 4. Use our existing query to pull the required data fields (i.e. Child first, middle, last name, DOB, City of birth, gender) to obtain the Global Unique Identifier (GUIDs).
  5. Descriptive/raw data will be submitted semi-annually (January and June); submission of all other data will be done at the time of publication and/or prior to the end of the grant. Positive and negative results will be shared. In addition to the NDCT, we are open to accepting requests for data use subsequent to publication of primary research findings.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At completion of study
Access Criteria: we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Stahmer AC, Lau AS, Roesch S, Rangel E, Aarons GA, Brookman-Frazee L. Understanding mechanisms of multi-level implementation strategies for autism interventions in a randomized trial across service systems. Implement Sci. 2025 Dec 15;20(1):54. doi: 10.1186/s13012-025-01466-z. PMID 41398285
- [Derived] Brookman-Frazee L, Lau AS, Roesch SC, Jobin A, Chlebowski C, Mello M, Caplan B, Naar S, Aarons GA, Stahmer AC. Effectiveness of Multilevel Implementation Strategies for Autism Interventions: Outcomes of Two Linked Implementation Trials. J Am Acad Child Adolesc Psychiatry. 2025 Dec;64(12):1386-1400. doi: 10.1016/j.jaac.2025.01.003. Epub 2025 Jan 13. PMID 39814315
- [Derived] Brookman-Frazee L, Stahmer AC. Effectiveness of a multi-level implementation strategy for ASD interventions: study protocol for two linked cluster randomized trials. Implement Sci. 2018 May 9;13(1):66. doi: 10.1186/s13012-018-0757-2. PMID 29743090
- See also: study website — https://www.teamsasdstudy.org/